CLINICAL TRIAL: NCT02970695
Title: Effectiveness of Auriculotherapy on Older People With Insomnia
Brief Title: Auriculotherapy on Older People With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Lorna Suen, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13144061
Record Dates: First submitted 2016-05-17; First posted 2016-11-22 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Insomnia
Keywords: insomnia; older people; auriculotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment arm 1 (Active Comparator): To achieve a blinding and placebo effect of the subject, the laser device will be switched to "power off" mode (i.e. deactivated laser) for acupoint "stimulation" before the application of MAT. The subjects will be asked to wear a pair of laser protective goggles so as to "blind" them during treatment.
  Interventions: Device: magneto-auriculotherapy (MAT)
- Treatment arm 2 (Active Comparator): Subjects will receive LAT. A laser device (Pointer Pulse™) will be used in this study.
  Interventions: Device: Laser auriculotherapy (LAT)
- Treatment arm 3 (Experimental): Subjects will receive a combined approach that includes the use of LAT plus MAT. LAT will be administered prior to MAT application on the selected auricular points, and the procedures used will be similar to the procedures described for Group 1 and Group 2.
  Interventions: Device: magneto-auriculotherapy (MAT); Device: Laser auriculotherapy (LAT)

INTERVENTIONS:
Device: magneto-auriculotherapy (MAT) — Subjects will then receive MAT. The magnetic pellets will have ~200 gauss/pellet magnetic flux densities on average, with a diameter of 1.76 mm.The experimental object will be applied to the seven selected acupoints as detected by an acupoint detector. Only one ear will receive treatment at a time, and the pellets will remain in situ for two days before the next change.
  Arms: Treatment arm 1; Treatment arm 3
Device: Laser auriculotherapy (LAT) — A laser device (Pointer Pulse™)15 will be used in this study. This device has a wavelength of 650 nm, an average output power of 2.5 mW, an energy density of 1 minute with 0.54 J/cm,2 and a pulse of 10 Hz, which is a common acceptable dosage for clinical use. 16, 17 This application is a low-energy laser therapy (LLLT), in which the energy level emitted from the device is approximately comparable to a teaching pointer. A 1-minute treatment using the continuous mode of the device will be directly applied to the selected acupoints. Laser protective goggles will be provided to the subjects and the researcher for eyes protection
  Arms: Treatment arm 2; Treatment arm 3

SUMMARY:
Objective To determine the optimum treatment protocol of auriculotherapy (AT) on the improvement of sleep conditions and quality of life on the elders with insomnia.

Research hypothesis The use of combined LAT plus MAT is more effective than MAT/LAT alone on the improvement of sleep conditions and quality of life in the elderly with insomnia.

Design and subjects This is a 3-arm double-blinded randomised trial. Subjects aged ≥65 and exhibit poor sleep conditions are recruited.

Interventions Group 1: Subjects will receive a deactivated laser treatment followed by MAT. Group 2: Subjects will receive LAT and placebo MAT. Group 3: Subjects will receive a combined approach (LAT plus MAT).

The treatment will be delivered 3 times/week, with a 6-week treatment period, on seven specific auricular points.

Main outcome measures Sleep conditions and quality of life will be evaluated at baseline; end of 6-week treatment; and at 6-week, 12-week, and 6-month follow-up periods.

Data analysis Descriptive statistics, chi-square analysis, ANOVA, paired t-test, and mixed effect modeling will be conducted as appropriate.

Expected results This study would advance our knowledge the optimum treatment protocol of AT in the improvement of the sleep conditions of the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who are aged 65 or above
* Report having difficulty falling or staying asleep, and/or frequent nocturnal awakenings
* At least three nights per week, sleep disturbance has lasted for a minimum of six months
* Their sleep is of poor quality as indicated by a PSQI score greater than five.

Exclusion Criteria:

* profound physical illness, such as stroke
* diagnosed with obstructive sleep apnoea
* having a hearing aid or pacemaker in situ (to prevent the magnetic pellets from interfering with the devices)
* receiving AT within the preceding 6 months,
* suffering from aural injuries or infections, and
* inability to understand instructions or give consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | up to 6-month follow up
  for collecting data related to the sleep patterns of the subjects. The total score ranges from 0 to 21, with a score greater than five indicating poor sleep quality. Chong and Cheung19 have validated the Cantonese-PSQI and have reported a high internal consistency of 0.75.

SECONDARY OUTCOMES:
Sleep latency | up to 6-month follow up
  Actiwatch 2 Device with 0.025G ultra-high sensitivity will be used for data collection. Sleep parameters, including sleep latency, waking after sleep onset, total sleep time, and sleep efficiency are identified. Participants have to wear the device for 7 consecutive days, 24 hours a day, for each timepoint measurements on the wrist of the non-dominant hand to determine the overall sleep conditions within a certain period. Removal (if any) of the actiwatch should be recorded in a logbook. Sleep latency refers to the length of time it takes from lying down for the night until sleep onset.
Wake after sleep onset | up to 6-month follow up
  Actiwatch 2 Device with 0.025G ultra-high sensitivity will be used for data collection. Sleep parameters, including sleep latency, waking after sleep onset, total sleep time, and sleep efficiency are identified. Participants have to wear the device for 7 consecutive days, 24 hours a day, for each timepoint measurements on the wrist of the non-dominant hand to determine the overall sleep conditions within a certain period. Removal (if any) of the actiwatch should be recorded in a logbook. Wake after sleep onset refers to the amount of time test subjects have spent awake after initially falling asleep and before they awaken for good.
Total sleep time | up to 6-month follow up
  Actiwatch 2 Device with 0.025G ultra-high sensitivity will be used for data collection. Sleep parameters, including sleep latency, waking after sleep onset, total sleep time, and sleep efficiency are identified. Participants have to wear the device for 7 consecutive days, 24 hours a day, for each timepoint measurements on the wrist of the non-dominant hand to determine the overall sleep conditions within a certain period. Removal (if any) of the actiwatch should be recorded in a logbook. Total sleep time refers to the actual sleep time in a sleep episode.
Sleep efficiency | up to 6-month follow up
  Actiwatch 2 Device with 0.025G ultra-high sensitivity will be used for data collection. Sleep parameters, including sleep latency, waking after sleep onset, total sleep time, and sleep efficiency are identified. Participants have to wear the device for 7 consecutive days, 24 hours a day, for each timepoint measurements on the wrist of the non-dominant hand to determine the overall sleep conditions within a certain period. Removal (if any) of the actiwatch should be recorded in a logbook. Sleep efficiency is the ratio of total time spent asleep (total sleep time) in an evening to the total amount of time spent in bed.
The Chinese (HK) specific SF-12 v2© | up to 6-month follow up
  to evaluate the quality of life of the subjects, and has been found to have positive psychometric properties for use in the local population
Patient Health Questionnaire | up to 6-month follow up
  to evaluate the depression status
Insomnia Severity Index | up to 6-month follow up
  to evaluate sleep conditions

OTHER OUTCOMES:
The 'Subjects' expectation questionnaire' | up to post-intervention at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Suen, BN, MPH, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- The Neighbourhood Advice-Action Council, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suen LKP, Molassiotis A, Yueng SKW, Yeh CH. Comparison of Magnetic Auriculotherapy, Laser Auriculotherapy and Their Combination for Treatment of Insomnia in the Elderly: A Double-Blinded Randomised Trial. Evid Based Complement Alternat Med. 2019 May 21;2019:3651268. doi: 10.1155/2019/3651268. eCollection 2019. PMID 31239857